CLINICAL TRIAL: NCT00862628
Title: The Effect of Rebamipide for Non-steroidal Anti-inflammatory Drugs (NSAID) - Induced Small-intestinal Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nagoya University (Other)
Responsible Party: Department of Gastroenterology, Nagoya University Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NO-003
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: NSAIDs-induced Small-intestinal Injuries
MeSH Terms: interventions — rebamipide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (1):
- Rebamipide (Experimental)
  Interventions: Drug: Rebamipide

INTERVENTIONS:
Drug: Rebamipide — 100mg tid, 4 or 8 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy of rebamipide for NSAID-induced small-intestinal injuries.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* 20 to 85 years of age
* RA, OA, or low back pain
* No change of drugs before 3 months
* Under 5 mg of corticosteroid use
* CRP < 1mg/dl
* Small-intestinal mucosal injuries more than one
* Hemoglobin level is below normal range

Exclusion Criteria:

* Known or suspected small-bowel disease, including Crohn's disease and seronegative arthritis
* Prostaglandins, metronidazole or salazosulfapyridine
* Can not swallow
* Eith pacemaker
* After gastrointestinal operation
* Serious concomitant cardiovascular, endocrine, gastrointestinal(including symptoms of ileus), neurologic, psychiatric, renal, or respiratory disease.
* Taking rebamipide before one week
* Any other conditions that the investigator feels would interfere with data interpretation or create under risk.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-06 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
The number of mucosal breaks | 4 and 8 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Ohmiya, M.D., Ph.D., Principal Investigator — Nagoya University Hospital
Locations (1):
- Department of Gastroenterology, Nagoya University Graduate School of Medicine, Nagoya, Aichi-ken, Japan